### **OMIT: STATISTICAL ANALYSIS PLAN**

Study Name: Calories or Time Restriction to Alter Biomarkers of Aging and Diabetes (OMIT)

Trial registration number(s): NCT05769335, H-2022-199

SAP Author: Andrew Vincent

**Signatures** 

Andrew Vincent (Senior Statistician, University of Adelaide) Andrew Vincent (Dec 20

Leonie Heilbronn (CI Lead, University of Adelaide)

Amy Hutchison (University of Adelaide) Amy Hutchison (Dec 20, 2024 10:02 GMT+10.5)

SAP Version: 1.0

SAP Date: 2024-12-19

SAP Revisions: None.

Protocol version used for SAP: Version 5 (approved 22/02/2024)

#### **CONTENTS**

Abbreviations (page 3)

Preface (page 4)

Study Objectives (page 5)

- Primary
- Secondary
- Exploratory

### Study Outcomes (page 6)

- Primary outcomes
- Secondary outcomes
- Exploratory outcomes

## Study Details (page 7)

- Study design
- Figure 1: Schedule of assessments
- Study Population: Inclusion/exclusion criteria
- Sample size considerations
- Randomization details

### Statistical Considerations (page 11)

- Estimand details
- Error control
- Covariate adjustment
- Sensitivity analyses

### Statistical Methods (page 14)

- Primary outcome
- Secondary outcomes
- Exploratory outcomes
- Safety outcomes

### Study Summary Tables (page 15)

- Descriptive statistics
- CONSORT diagram

# References (page 16)

Appendix: Results summary tables (page 17)

Code for imputation (R) (page 23)

# **ABBREVIATIONS**

| AUC | Area under the curve |
|----------|-------------------------------------------------------------------|
| AUSDRISK | The Australian type 2 diabetes risk assessment tool |
| BMI | Body mass index |
| CGM | Continuous glucose monitoring |
| CR | Calorie restriction (30%) |
| dCR | Delayed calorie restriction (30% calorie restriction, 12pm – 8pm) |
| eCR | Early calorie restriction (30% calorie restriction, 8am – 4pm) |
| HbA1c | Glycated haemoglobin |
| iAUC | Incremental area under the curve |
| PP | Post-prandial |
| SAP | Statistical analysis plan |
| T2DM | Type II diabetes mellitus |

### **PREFACE**

This statistical analysis plan (SAP) describes the planned analyses and reporting for the OMIT study to compare early calorie restriction (eCR) or delayed calorie restriction (dCR) versus calorie restriction (CR) without time limits in men and women with overweight and obesity and elevated fasting blood glucose. The purpose of this SAP is to outline the considerations and the pre-specified analyses for the OMIT study.

The project is funded by the NHMRC Ideas grant #2012569 awarded to Prof Leonie Heilbronn.

This study has been approved by the University of Adelaide Human Research Ethics Committee (HREC 2022-199).

### **Study Rationale & Objectives**

### Background/Rationale

Caloric restriction (CR) is widely recognised for its ability to reverse or alleviate the metabolic health consequences of obesity, and even extends lifespan in mouse models. Time-restricted eating (TRE), whereby food intake is typically limited to 8 h eating window during the day may be a novel, alternative dietary strategy to improve cardiometabolic health individuals with obesity. Recent studies in mice suggest that CR+TRE was able to extend the health benefits of CR alone, with the maximal effect noted when the meal timing period was initiated at the onset of the active phase. The ideal meal timing to initiate TRE is under-researched in humans. The proposed randomised clinical trial will be the first to determine whether CR+TRE that is initiated early in the day (early CR) or delayed CR is able to extend the health benefits of CR alone in humans.

### **Primary Objective**

- To establish whether early or delayed time-restricted eating plus calorie restriction, improve markers of type 2 diabetes, compared with calorie restriction alone.

### **Secondary Objective**

- To explore the effect of time-restricted eating on insulin and gut peptide AUCs, 24-h glycaemia by CGM, and cardiometabolic health biomarkers.

#### **Study Outcomes**

### **Primary efficacy outcomes**

- The difference in percentage change from baseline in the mean 2-hour post-meal glucose AUC levels after eight weeks of (i) time restricted (early) versus non-time restricted dieting and (ii) time restricted (delayed) versus non-time restricted dieting, in men and women with obesity.

### Secondary efficacy outcomes at 8 weeks

- Changes in...
  - o PP insulin AUC
  - o fasting insulin,
  - o fasting glucose, and
  - o HbA1c.

### **Exploratory mechanistic outcomes:** at 8 weeks

- Change in...
  - o PP glucose and insulin AUCs for each meal
  - 24-h glucose by CGM (mean and iAUC),
  - nocturnal glucose by CGM (mean)
  - o insulin sensitivity calculated by the Matsuda index
  - gut peptides (AUCs and iAUC),
  - o insulin secretion by C-peptide,
  - o HOMA-IR
  - 24-h profiles of glycaemia by CGM (i.e. time-above/below/in range, MAGE, MODD)

### **Exploratory outcomes**

- Listed in the Appendix, see tables A4 & A5.

#### **Compliance outcomes**

- Self-reported adherence over the eight weeks
- Adherence to eating window assessed by smartphone application and diet diaries.
- Protocol deviations arising from inappropriate inclusion (ie contradicting inclusions/exclusion criteria) will be listed.

# **STUDY DETAILS**

**Study Design:** OMIT is a three-arm parallel, single-blinded, single-centre randomised controlled clinical trial.

Figure 1: Schedule of assessments



### **Study Population**

#### Inclusion criteria

Study participants will be aged 35 to 75 years and overweight (BMI: >25.1 but < 45kg/m2) with elevated waist circumference, score 12 or greater on the AUSDRISK questionnaire and have elevated fasting blood glucose (≥5.6 mmol/L).

| Elevated risk for waist circumference | Male(cm) | Female (cm) |
|------------------------------------------------|----------|-------------|
| Caucasian/African | >94 | >80 |
| Asian | >88 | >74 |
| South Asian, Aboriginal/Torres Strait Islander | >79 | >70 |

#### Exclusion criteria

A personal history/diagnosis (self-reported) of:

- diabetes (type 1 or 2)
- major psychiatric disorders (schizophrenia, major depressive disorder, bipolar disorder, eating disorders)
- gastrointestinal disorders/disease (including malabsorption)
- haematological disorders (i.e. thalassemia, iron-deficiency anaemia)
- insomnia
- obstructive sleep apnea
- night eating syndrome
- currently receiving, or have received treatment/diagnosis of cancer in the past 3 years (excluding non-melanoma skin cancer)
- significant liver or kidney diseases that require ongoing medical care
- previous or planned gastro-intestinal surgery (including bariatric surgery)
- Congestive heart failure (NYHA stage 2 or above)
- Previous myocardial infarction or significant cardiac event ≤ 6 months prior to screening
- Previous cerebrovascular event ≤ 12 months prior to screening
- Any autoimmune disease (i.e. rheumatoid arthritis)
- Coeliac disease/gluten allergy
- Nut allergy
- other conditions deemed unstable by the study physician.

### Currently taking the following medications:

- used, or known, to lower blood glucose, or antidiabetic medications, including, but not limited to: SGLT2 inhibitors, metformin, sulfonylureas, glucagon-like peptide-1 analogues [i.e. exenatide], thiazolidinediones or DPP-IV inhibitors [i.e. 'gliptins'])
- affecting weight, appetite or gut motility, including, but not limited to: (domperidone, cisapride, orlistat, phentermine, topiramate).
- Diuretics (i.e. thiazides) or combination blood pressure medications containing a

#### diuretic

- Beta-blockers
- Glucocorticoids
- Anti-epileptic medications (i.e. pregabalin and gabapentin)
- Tricyclic antidepressants
- Some serotonin and norepinephrine reuptake inhibitors (i.e. vortioxetine, mirtazapine and venlafaxine)
- Regular use of benzodiazepines or other sleep aids, including melatonin
- Antipsychotic medications
- Opioid medications unless combined with paracetamol in a single formulation and used occasionally on a PRN basis

Participants who are taking stable doses (i.e. > 3 mo.) of androgenic medications (i.e. testosterone), blood pressure medications (not listed above), lipid medications, thyroid medication, SSRI's or SNRIs (with the exception of those mentioned above) or benign prostatic hyperplasia will not be excluded.

#### Additional exclusion criteria include:

- AUSDRISK score of < 12
- Fasting blood glucose levels < 5.6
- Score ≥ 30 on Kessler Psychological Distress scale
- do not eat for 12 hours per day on an average of 5 or more days per week
- have extreme or restricted patterns of eating (i.e. following an intermittent fasting diet) or already engage in CR or TR
- night shift-workers (>3 shifts per month)
- pregnant, planning a pregnancy or currently breastfeeding
- those who have lost or gained >5% of body weight in the last 6 months
- donated blood in past 3 months
- current smokers of cigarettes/marijuana/e-cigarettes/vaporisers
- anyone unable to comprehend the study protocol or provide informed consent (i.e. due to English language or cognitive difficulties)
- do not own, or are not comfortable using, a smartphone and applications

Individuals with dietary restrictions or practices, including vegans and those with gluten or nut allergies will be excluded. Less restrictive dietary practices including vegetarians and those with lactose intolerance or specific dietary dislikes will be accommodated.

### **Pre-planned Sample size**

An expected group difference is 0.46 mmol/L at 2-hrs after a glucose tolerance test (1). Our past data, DIRECT study (2) showed a mean glucose concentration of 7 mmol/L at two hours post meal. We note that 0.46/7.0 is a 6.5% reduction. T4DM powered for a 0.6 mmol/L between group difference, which is approximatively 6% change from baseline in a population including individuals with diabetes (3). We thereby assumed the MCID to be a 6% reduction from baseline in mean post meal AUC and use log (AUC) to estimate of the percentage difference between groups (4).

Using data from the DIRECT study (2), the SD of the log (meal test AUC) is expected to be 0.152 and pre-post AUC correlations were 0.87 at breakfast and 0.92 at dinner.

With N=114 (38 per group, randomized 1:1:1), a within-group SD of 0.152, pre-post correlation of at least 0.85 and a drop-out rate less than 10%, there is >80% to detect a difference of 0.06 in log-transformed AUC in a baseline adjusted ANCOVA (alpha = 0.027 two-sided) (5).

### Sample size adaption

None

#### Randomization details

Stratified random length blocked randomisation by sex (male or female) and fasting plasma glucose ( $\leq$ 6.0 vs >6.0 mmol/L)

### **STATISTICAL CONSIDERATIONS**

### **Estimand Considerations**

### Study objective

- To establish whether early or delayed time-restricted eating plus calorie restriction (eCR, dCR), improve markers of type 2 diabetes, compared with calorie restriction (CR) alone

### **Estimand**

- The difference in percentage change from baseline in the mean 2-hour post-meal glucose AUC levels after eight weeks of time restricted versus non-time restricted dieting, in obese men and women

#### **Treatment**

- eCR (30% calorie restriction, 8am 4pm);
- dCR (30% calorie restriction, 12pm 8pm);
- CR (30% calorie restriction, 8am-8pm); Control group

| ESTIMA | AND | ANALY | SIS |
|---|---|---|---|
| Target | population | Analysi | is set |
| - | Men and women with obesity and | - | All randomized |
| | elevated fasting blood glucose | - | Initiated diet |
| Variab | le | Outcor | ne measure |
| - | Glucose AUC over 3 meals (breakfast, | - | Blood glucose AUC |
| | lunch, dinner). | - | Measured at 0,30,60,120 post-meal |
| | | - | Averaged over three meals |
| Handli | ng of inter-current events | | ng of missing data |
| 1. | Death (while on treatment strategy, | 1. | Death believed not to be relevant |
| | or "while alive") | | for this study, included for |
| 2. | Discontinuation: other reason (while | | completeness. |
| | on treatment strategy) | 2. | All individuals discontinuing early |
| 3. | Discontinuation: dislike of diet | | will (i) be invited to attend the week |
| | (treatment policy strategy) | | 6 assessment for fasting bloods and |
| 4. | Lost-to-follow-up no reason | | body weight only, (ii) asked whether |
| | provided (treatment policy strategy) | | the reason for discontinuation is |
| | | | due to allocated diet. |
| | | 3. | Missing-at-random will be assumed |
| | | | for individuals who do not specify |
| | | | whether discontinuation was due to |
| | | | diet, or when the reason was not due to the diet. |
| | | 4 | For individuals who discontinued |
| | | 4. | due to the diet a missing-not-at- |
| | | | random assumption will be made, |
| | | | assuming zero adherence after |
| | | | discontinuation, and conditional on |
| | | | adherence missing-at-random |
| | | | assumed to impute week 8 |
| | | | outcomes. |
| | | I | |

#### 5. Imputation is by treatment group with individuals imputed in the groups they were allocated to. Population level summary measure **Analysis approach** Mean between group differences in Group differences of log baseline adjusted log-transformed transformed mean post-prandial (within-individual) mean post-meal AUC will be estimated using a single glucose AUC, of the time-restricted linear regression with a treatment groups verses the control (non time-(three levels) and baseline log restricted) group. transformed mean post-prandial glucose AUC and stratification factors (sex and fasting plasma glucose).

**Hypothesis testing framework:** All analyses are to test for superiority of eCR and dCR over CR.

**Analyses:** No interim analyses are planned. The analysis of the primary outcome will be conducted after the final subject has completed their 8 week assessment and the blood samples assessed for glucose concentrations.

**Error Control:** There are two primary comparisons, eCR vs CR and dCR vs CR with a common control and thereby use a Dunnett multi-test adjustment that controls the familywise error rate at 0.05 (two-sided) when each pairwise test uses an alpha of 0.027 (two-sided).

There are four secondary efficacy outcomes that will be tested to support a confirmatory finding: (i) PP insulin AUC, (ii) fasting insulin, (iii) fasting glucose, and (iv) HbA1c. An ordered testing procedure with per comparison (eCR vs CR and dCR vs CR) will be applied testing these four secondary outcomes in the order listed here, testing each subsequent outcome only if the previous outcome (and primary outcome) rejected the null. This procedure is applied separately for each comparison: eCR vs CR and dCR vs CR. The same pairwise alpha level, 0.027 (two sided), as the primary outcome will be applied to ensure that the familywise error rate is controlled at 0.05 (two-sided).

Standard multiplicity unadjusted 95% confidence intervals will be reported for all comparisons.

Covariate adjustment: All comparisons of treatment effect will include adjustment for...

- 1. The outcome variable's baseline assessment if appropriate,
- 2. Stratification factors (sex and baseline fasting plasma glucose as a continuous variable)

**Sensitivity Analyses:** A best-worst case sensitivity analysis will be performed for the analysis of the primary outcome and secondary efficacy outcomes.

- For all individuals missing the week 8 assessment in the CR (control) group the outcome will be imputed assuming missing-at-random. In other words, as if each individual's mean adherence was continued, or the cohort's mean adherence if no adherence data is available for an individual.
- For individuals in missing the week 8 assessment in the eCR and dCR groups their outcome, a missing-not-at-random assumption will be applied by assuming zero adherence and outcomes imputed thereafter, i.e., assuming missing-at-random conditional on zero subsequent adherence.
- These assumptions will be made irrespective of the stated reason for diet discontinuation.

A secondary, complete-case sensitivity analysis will be performed for the analysis of the primary outcome and secondary efficacy outcomes in this analysis individuals with both baseline and week 8 assessments will only be included for each analysis.

As additional analysis will explore the treatment effects within subjects who were adherent to the protocol using data collected with the MyCircadianClock app plus the dietary checklists. This analysis will be reported in a secondary mechanistic publication of this study.

### **STATISTICAL METHODS**

#### **Primary Outcome**

The primary analysis of the primary outcome is a covariate adjusted linear regression of the differences in PP glucose log AUC at 8 weeks from baseline. Covariates included will be treatment (three groups), baseline glucose log AUC, sex and fasting plasma blood glucose (as a continuous linear variable). Visual inspection of the residual distribution will be used to determine if assumptions of normality and the absence of a variance-mean association appear to be violated. If assumptions appear violated a generalized linear models will be considered with differing link functions will be considered and presented as sensitivity analyses. Given the limited sample size, no subgroup analyses are planned.

This analysis will be performed in all randomized individuals with individuals using multiple imputation using chained equations within treatment groups and combined using Rubin's rules. The variables used in the multiple imputation are age and sex; baseline and week 8 assessments of weight, PP glucose and insulin AUC (per meal), fasting glucose, fasting insulin and HbA1c; and the self-reported adherence over the 8 weeks and reason for discontinuation (related/unrelated to diet) if applicable. All concentrations will be imputed on the log scale, with the 3-meal mean of PP glucose and insulin AUC being calculated on the original scale after a back-transformation. Compliance will be imputed as per the intercurrent event strategies and the average compliance calculated over each period. Imputation will use multiple chained equations (*mice* R package), details of which are attached separately (file: *OMIT – Imputation code 2024-12-18.r*).

#### Secondary Efficacy Outcomes

The four secondary efficacy outcomes used in the multiple imputation of the primary outcome will be assessed using the same methodology as for the primary outcome, i.e. covariate adjusted linear regressions with multiple imputation for missing data.

#### **Exploratory Outcomes**

Exploratory outcomes will also be analysed using baseline and stratification factor adjusted linear regressions. The weight and PP glucose and insulin meal specific analyses will be performed in the imputed data sets. All other outcomes will be analysed using complete case data sets.

### Safety Outcomes

Summaries, for all adverse events and for those events believed to be related to the intervention, will be reported. In both cases, if an individual has experienced the adverse event on multiple occasions, only the event with the maximum grade will be reported.

When there are at least four individuals who experience a particular adverse event, a Fisher exact test will be conducted comparing the rates of occurrence (irrespective of grade) between the two intervention groups. No adjustments for multiple testing will be performed.

### **STUDY SUMMARY TABLES**

**Descriptive Statistics:** A CONSORT flow chart will present all individuals screened through to randomization and week 8 assessment will be presented (Figure 2). The number of individuals who discontinue their allocated intervention and/or withdraw from the study, the week and reason for discontinuation will be reported.

Descriptive summary statistics will be reported for baseline characteristics of all individuals who were randomized. In addition to baseline glycemia indices we will report on age, sex, menopausal status, AUSDRISK, body composition, markers of CVD risk, sleep, activity and appetite measures. For continuous variables means, standard deviations, medians and ranges will be reported, and for discrete variables frequency and percentages will be reported. No demographic summary statistics were collected for the screened cohort.

Results tables presenting the analyses of the primary, secondary and exploratory outcomes are presented in Appendix A.

Figure 2: CONSORT flow chart of OMIT study.



#### **REFERENCES**

- 1. Hemmingsen B, Gimenez-Perez G, Mauricio D, Roqué I Figuls M, Metzendorf MI, Richter B. Diet, physical activity or both for prevention or delay of type 2 diabetes mellitus and its associated complications in people at increased risk of developing type 2 diabetes mellitus. Cochrane Database Syst Rev. 2017 Dec 4;12(12):CD003054.
- 2: Teong XT, Liu K, Vincent AD, Bensalem J, Liu B, Hattersley KJ, Zhao L, Feinle-Bisset C, Sargeant TJ, Wittert GA, Hutchison AT, Heilbronn LK. Intermittent fasting plus early time-restricted eating versus calorie restriction and standard care in adults at risk of type 2 diabetes: a randomized controlled trial. Nat Med. 2023 Apr;29(4):963-972. doi: 10.1038/s41591-023-02287-7. Epub 2023 Apr 6. PMID: 37024596.
- 3. Wittert G, Bracken K, Robledo KP, Grossmann M, Yeap BB, Handelsman DJ, Stuckey B, Conway A, Inder W, McLachlan R, Allan C, Jesudason D, Fui MNT, Hague W, Jenkins A, Daniel M, Gebski V, Keech A. Testosterone treatment to prevent or revert type 2 diabetes in men enrolled in a lifestyle programme (T4DM): a randomised, double-blind, placebo-controlled, 2-year, phase 3b trial. Lancet Diabetes Endocrinol. 2021 Jan;9(1):32-45.
- 4. Cole TJ. "Sympercents: symmetric percentage differences on the 100loge scale simplify the presentation of log transformed data." Statistics in medicine 2000; 19: 3109-3125.
- 5. Borm GF, Fransen J, Lemmens WA. A simple sample size formula for analysis of covariance in randomized clinical trials. J Clin Epidemiol. 2007 Dec;60(12):1234-8

# **Appendix A: Results Tables.**

**Table A1**: Primary outcome and confirmatory secondary outcomes with ordered testing procedure per comparison. Analyses from the prespecified multiply imputed analysis.

| | A: Est [95% CI] | B: Est [95% CI] | C: Est [95% CI] | AvC: Est [95% CI] | AvC p-value | BvC: Est [95% CI] | BvC p-value |
|---|---|---|---|---|---|---|---|
| PP glucose AUC | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| PP insulin AUC | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | * | NA [NA; NA] | * |
| Fasting insulin | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | * | NA [NA; NA] | * |
| Fasting glucose | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | * | NA [NA; NA] | * |
| HbA1c | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | * | NA [NA; NA] | * |

**Table A2**: Best-worst case sensitivity analysis of the primary analysis.

| | A: Est [95% CI] | B: Est [95% CI] | C: Est [95% CI] | AvC: Est [95% CI] | BvC: Est [95% CI] |
|---|---|---|---|---|---|
| PP glucose AUC | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] |
| PP insulin AUC | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] |
| Fasting insulin | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] |
| Fasting glucose | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] |
| HbA1c | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] |

**Table A3**: Complete case sensitivity analysis of the primary analysis.

| | A: Est [95% CI] | B: Est [95% CI] | C: Est [95% CI] | AvC: Est [95% CI] | BvC: Est [95% CI] |
|---|---|---|---|---|---|
| PP glucose AUC | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] |
| PP insulin AUC | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] |
| Fasting insulin | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] |
| Fasting glucose | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] |
| HbA1c | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] |

**Table A4**: Exploratory outcome analyses for outcomes used in the multiple imputation of the primary outcome, ie using the imputed data.

| | A: Est [95% CI] | B: Est [95% CI] | C: Est [95% CI] | AvC: Est [95% CI] | AvC p-value | BvC: Est [95% CI] | BvC p-value |
|---|---|---|---|---|---|---|---|
| Glucose.auc.break | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Glucose.auc.lunch | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Glucose.auc.dinner | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Insulin.auc.break | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Insulin.auc.lunch | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Insulin.auc.dinner | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Weight | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |

**Table A5**: Exploratory outcome analyses for outcomes not used in the multiple imputation of the primary outcome, ie complete case analyses.

| | A: Est [95% CI] | B: Est [95% CI] | C: Est [95% CI] | AvC: Est [95% CI] | AvC p-value | BvC: Est [95% CI] | BvC p-value |
|---|---|---|---|---|---|---|---|
| Mean Glucose CGM | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| iAUC glucose CGM | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Nocturnal glucose CGM | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| CGM time below range | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| CGM time in range | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| CGM time above range | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| MAGE | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| MODD | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Insulin secretion rate | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Insulin sensitivity index | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| HOMA-IR | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Fasting C-peptide | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Fasting Triglycerides | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Fasting free fatty acids | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Trigs AUC of 3 meals | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Trigs AUC of breakfast | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Trigs AUC of lunch | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Trigs AUC of dinner | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| FFA AUC of 3 meals | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| FFA AUC of breakfast | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |

| FFA AUC of lunch | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
|---|---|---|---|---|---|---|---|
| FFA AUC of dinner | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Systolic BP | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Diastolic BP | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Total cholesterol | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| HDL | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| LDL | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| C-reactive protein | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| ВМІ | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Sleep duration | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Arousals | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| AHI | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Light sleep | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Deep sleep | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| REM sleep | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Sleep latency | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Sitting time | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Standing time | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Stepping time | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Mean daily steps | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Adherence | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Eating window | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| 95% Eating window | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Protein | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Carbohydrate | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Fat | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Sat fat | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Fibre | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Alcohol | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Hunger AUC 3 meals | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Hunger AUC breakfast | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Hunger AUC lunch | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Hunger AUC dinner | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Fullness AUC 3 meals | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Fullness AUC breakfast | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Fullness AUC lunch | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| • | | | | | | | |

| Fullness AUC dinner | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
|---|---|---|---|---|---|---|---|
| Desire AUC 3 meals | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Desire AUC breakfast | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Desire AUC lunch | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Desire AUC dinner | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Consumption AUC 3 meals | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Consumption AUC breakfast | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Consumption AUC lunch | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Consumption AUC dinner | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Fasting ghrelin | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Ghrelin AUC of 3 meals | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Ghrelin AUC of breakfast | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Ghrelin AUC of lunch | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Ghrelin AUC of dinner | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| Fasting GLP1 | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| GLP1 AUC of 3 meals | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| GLP1 AUC of breakfast | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| GLP1 AUC of lunch | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |
| GLP1 AUC of dinner | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA [NA; NA] | NA | NA [NA; NA] | NA |

# Appendix B: SAP checklist.

| Section | Index | Page | Description |
|---|---|---|---|
| 1: Administration | 1a | 1 | Title matches the protocol with SAP as forerunner or subtitle |
| | 1b | 1 | Trial registration number |
| | 2 | 1 | SAP version number with dates |
| | 3 | 1 | Reference to version of protocol being used |
| | 4a | 1 | SAP revision history |
| | 4b | NA | Justification for each revision |
| | 4c | NA | Timing of SAP revisions in relation to interim analyses |
| | 5 | 1 | Names, affiliations and roles of SAP contributors |
| | 6a | 1 | Person writing SAP |
| | 6b | 1 | Senior statistician responsibility |
| | 6c | 1 | Chief investigator/Clinical lead |
| 2: Introduction | 7 | 5 | Synopsis of trial background and rationale |
| | 8 | 5 | Description of specific objectives or hypothesis |
| 3: Study Methods | 9 | 7 | Brief description of trial design |
| | 10 | 10 | Randomisation details |
| | 11 | 10 | Sample size calcs |
| | 12 | 12 | Superiority/equiv/non-inferiority |
| | 13a | 12 | Info regarding interim analyses |
| | 13b | NA | Adjustment to significance |
| | 13c | NA | Stopping rules |
| | 14 | 12 | Timing of final analysis |
| | 15 | 6 | Time points at which outcomes are measured |
| 4: Statistical principals | 16 | 12 | Level of statistical significance |
| | 17 | 12 | Rationale for multiplicity adjustments and T1 error control |
| | 18 | 12 | Confidence intervals to be reported. |
| | 19a | 6 | Definition of adherence |
| | 19b | 6 | Description of how adherence will be presented |
| | 19c | 6, 8, 9 | Definition of protocol deviations |

| | 19d | 6 | Description of which deviations will be summarized |
|---|---|---|---|
| | 20 | 11 | Definition of analysis populations |
| 5: Trial population | 21 | 15 | Reporting of screening data to describe representativeness of trial sample |
| | 22 | 8,9 | Summary of eligibility criteria |
| | 23 | 15 | Information to be included in CONSORT flow chart |
| | 24a | 15 | Level of withdrawal, from intervention and/or follow-up |
| | 24b | 15 | Timing of withdrawals |
| | 24c | 15 | Reasons and details how withdrawals will be presented. |
| | 25a | 15 | List of baseline characteristics to be summarized |
| | 25b | 15 | Details of how baseline characteristics will be summarized |
| 6: Analysis | 26 | 6 | List of primary and secondary outcomes |
| | 26a | 12 | Outcome timings and order of importance |
| | 26b | 10, 11 | Specific measurement and units |
| | 26c | 14 | Calculation or transformation used to derive the outcome |
| | 27a | 14 | Analysis method to estimate treatment effects |
| | 27b | 12 | Covariates adjusted for |
| | 27c | 14 | Methods to check assumptions |
| | 27d | 14 | Details of alternative methods if distributional assumptions do not hold |
| | 27e | 13 | Planned sensitivity analyses |
| | 27f | 14 | Planned subgroup analyses and definitions of subgroups |
| | 28 | 11, 12 | Assumptions methods for dealing with missing data. |

# OMIT STUDY – CODE FOR IMPUTATION (R) 18-12-2024





```
for (visit. in c('w0', 'w8')) {
  imp.data[,paste(var., visit., sep='.')] <- log(imp.data[,paste(var., visit., sep='.')])</pre>
 }; rm(visit.)
}; rm(var.)
## Variable lists
w0.list <- names(imp.data)[grepl('w0', names(imp.data))]
sum(!w0.list %in% names(imp.data)) # 0
w0.list <- w0.list[order(colSums(is.na(imp.data[,w0.list])))]; w0.list
w8.list <- names(imp.data)[grepl('w8', names(imp.data)) & !grepl('adher', names(imp.data))]
```

```
sum(!w8.list %in% names(imp.data)) # 0
w8.list <- w8.list[order(colSums(is.na(imp.data[,w8.list])))]; w8.list
calculated.list <- c("adherence", "glucose.auc.w0", "insulin.auc.w0", "glucose.auc.w8", "insulin.auc.w8")
w0.list <- w0.list[!w0.list %in% calculated.list]
w8.list <- w8.list[!w8.list %in% calculated.list]
adher.list <- c('drop.out', 'week.drop', 'adher.w2', 'adher.w4', 'adher.w8')
sum(!adher.list %in% names(imp.data)) # 0
aux.list <- c("id", "treat", 'sex');</pre>
```

sum(!aux.list %in% names(imp.data)) # 0 table(table(c(w0.list, w8.list, aux.list, adher.list, calculated.list))) # all 1s sum(!names(imp.data) %in% c(w0.list, w8.list, aux.list, adher.list, calculated.list)) # 0 ## List of meal data for formula construction meal.list <- c( "glucose.auc.break.w0", "glucose.auc.lunch.w0", "glucose.auc.dinner.w0" , "insulin.auc.break.w0", "insulin.auc.lunch.w0", "insulin.auc.dinner.w0" , "glucose.auc.break.w8", "glucose.auc.lunch.w8", "glucose.auc.dinner.w8"

, "insulin.auc.break.w8", "insulin.auc.lunch.w8", "insulin.auc.dinner.w8"

```
sum(!meal.list %in% names(imp.data)) # 0
###################
## Multiple Imputation
#####################
## MI
set.seed(1234)
M. <- 100; N.iter <- 100
```

```
options(warn=0)
time. <- Sys.time()
for (MNAR.type in 0:1) {
 ## Code assumes control group = 'C'
 library(mice)
 # Set up data assumptions dropout
  temp.data <- imp.data[, c(w0.list, w8.list, calculated.list, aux.list, adher.list)]
  colSums(is.na(temp.data))
```

```
## MAR: impute unknown drop out reason.
if (MNAR.type == 0) {
 temp.data$drop.out[temp.data$drop.out == 'Unknown'] <- NA
 sum(length(unique(temp.data$drop.out)) != 3) # 0
## MNAR: Do not impute unknown drop.out, set at best-worst case: A & B due to diet vs C not diet
if (MNAR.type == 1) {
 temp.data$drop.out[temp.data$treat == 'C' & temp.data$drop.out == 'Unknown'] <- 'Not diet'
 temp.data$drop.out[temp.data$treat %in% c('A', 'B') & temp.data$drop.out == 'Unknown'] <- 'Diet'
 sum(length(unique(temp.data$drop.out)) != 3) # 0
```

```
temp.data$drop.out <- temp.data$drop.out[drop=T]
if (nlevels(temp.data$drop.out) != 2) cat('Error wrong number of drop options.\n')
## Set individuals who did not discontinue to 'Not diet' drop out at week 8 (ie so data is not imputed)
cond. <- rowSums(!is.na(temp.data[,w8.list[w8.list != 'fasting.glucose.w8']])) > 0
temp.data$drop.out[is.na(temp.data$drop.out) & cond.] <- 'Not diet'
temp.data$week.drop[is.na(temp.data$week.drop) & cond.] <- 8; rm(cond.)
## Set adherence to "Strongly Disagree" (ie 0) when due to diet and after drop-out week
for (id. in temp.data$id[temp.data$drop.out == 'Diet' & !is.na(temp.data$drop.out)]) {
```

```
week. <- temp.data$week.drop[temp.data$id == id.]</pre>
 if (week. < 2) temp.data$adher.w2[temp.data$id == id.] <- 0
 if (week. < 4) temp.data$adher.w4[temp.data$id == id.] <- 0
 if (week. < 8) temp.data$adher.w8[temp.data$id == id.] <- 0
 rm(week.)
}; rm(id.)
## Calculate mean adherence over the eight weeks.
temp.data$adherence <- ((temp.data$adher.w2) + (temp.data$adher.w4) + 2*(temp.data$adher.w8))/4
```

```
# Set up imputation functions
 fm.list <- NULL
 for (var. in w0.list) { # [!sub('.w0', ", w0.list) %in% data.list$log.list]
  if (!var. %in% meal.list) {
   fm. <- paste(var., "~ sex + ", paste(c(w0.list[!w0.list %in% c(var., meal.list)], "glucose.auc.w0", "insulin.auc.w0"), collapse=' + '))
   fm.list <- c(fm.list, as.formula(fm.)); rm(fm.)
  } else {
   fm. <- paste(var., "\sim sex + ", paste(c(w0.list[!w0.list %in% (var.)]), collapse=' + '))
   fm.list <- c(fm.list, as.formula(fm.)); rm(fm.)
```

```
}; rm(var.)
for (var. in w8.list) {
 # var. <- w8.list[1]
 if (!var. %in% meal.list) {
  fm. <- paste(var., "~ (", paste(c(
   sub('w8', 'w0', var.)
   , c('sex', 'adherence', "fasting.glucose.w0", "glucose.auc.w0", "insulin.auc.w0")
   , w8.list[!w8.list %in% c(var., meal.list)]
   , c("glucose.auc.w8", "insulin.auc.w8")
  ), collapse=' + '), ')')
  fm.list <- c(fm.list, as.formula(fm.)); rm(fm.)
```

```
} else {
  fm. <- paste(var., "~ (", paste(c(
   sub('w8', 'w0', var.)
   , c('sex', 'adherence', 'fasting.glucose.w0')
   , w8.list[!w8.list %in% c(var.)]
   ), collapse=' + '), ')')
   fm.list <- c(fm.list, as.formula(fm.)); rm(fm.)
}; rm(var.)
fm.list <- as.list(fm.list)
names(fm.list) <- c(w0.list, w8.list)
```

```
## Drop out & adherence
  fm.list$drop.out <- as.formula('drop.out ~ 1')
  fm.list$adher.w2 <- as.formula('adher.w2 ~ 0 + I(as.numeric(drop.out != "Diet")*as.numeric(week.drop >= 2))')
  fm.list$adher.w4 <- as.formula('adher.w4 ~ 0 + I(as.numeric(drop.out != "Diet")*as.numeric(week.drop >= 4)*as.numeric(adher.w2))')
  fm.list$adher.w8 <- as.formula('adher.w8 ~ 0 + I(as.numeric(drop.out != "Diet")*as.numeric(adher.w2)) + I(as.numeric(drop.out !=
"Diet")*as.numeric(adher.w4))')
 library(mice)
```
```
# Set up imputation methods
var.list <- c(w0.list, adher.list, w8.list, calculated.list)
 mice.fit <- mice(
  data=temp.data
  , m=1, maxit=0
  , blocks=var.list
  , visitSequent=var.list
  , formulas=fm.list
 mice.fit$loggedEvents
```

```
method. <- mice.fit$method
## Construct calculated methods
 method.[names(method.) == 'glucose.auc.w0'] <- gsub(
  '\n', '',
  "~ I(
   log((
    exp(glucose.auc.break.w0)
    + exp(glucose.auc.lunch.w0)
    + exp(glucose.auc.dinner.w0)
```

```
)/3)
 )"
method.[names(method.) == 'insulin.auc.w0'] <- gsub(
 '\n', '',
 "~ I(
  log((
   exp(insulin.auc.break.w0)
   + exp(insulin.auc.lunch.w0)
   + exp(insulin.auc.dinner.w0)
  )/3)
```

```
)"
method.[names(method.) == 'glucose.auc.w8'] <- gsub(
'\n', '',
"~ I(
  log((
   exp(glucose.auc.break.w8)
   + exp(glucose.auc.lunch.w8)
   + exp(glucose.auc.dinner.w8)
  )/3)
```

```
method.[names(method.) == 'insulin.auc.w8'] <- gsub(
 '\n', '',
 "~ I(
  log((
   exp(insulin.auc.break.w8)
   + exp(insulin.auc.lunch.w8)
   + exp(insulin.auc.dinner.w8)
  )/3)
 )"
```

```
method.[names(method.) == 'adherence'] <- gsub(
 '\n', '',
 "~ I(
  ((
   as.numeric(adher.w2)
   + as.numeric(adher.w4)
   + 2*as.numeric(adher.w8)
  )/4)
 )"
```

```
for (treat. in c('A', 'B', 'C')) {
 mice.fit2 <- mice(
  data=temp.data[temp.data$treat == treat.,]
  , m=M., maxit=N.iter
  , blocks=var.list
  , visitSequent=var.list
  , formulas=fm.list
  , method=method.
  , print=F
```

```
mice.fit2$loggedEvents
 if (treat. == 'A') mice.fit.A <- mice.fit2
 if (treat. == "B") mice.fit.B <- mice.fit2
 if (treat. == "C") mice.fit.C <- mice.fit2
 rm(mice.fit2)
}; rm(treat.)
rm(mice.fit, method., fm.list, var.list)
```



```
output <- NULL
for (MNAR.type in 0:1) {
 if (MNAR.type == 0) mice.full.fit <- mice.full.fit0
 if (MNAR.type == 1) mice.full.fit <- mice.full.fit1
 library(mice)
 var.list <- c(
  'glucose.auc', "glucose.auc.break", "glucose.auc.lunch", "glucose.auc.dinner", 'fasting.glucose'
  , 'insulin.auc', "insulin.auc.break", "insulin.auc.lunch", "insulin.auc.dinner", 'fasting.insulin'
  , 'weight', "hba1c"
```

```
for (var. in var.list) {
 for (visit. in c('.w8')) {
  output <- rbind(output, c(</pre>
   c('MI', 'MI-worst')[0:1 == MNAR.type]
   , 'diff - orig'
   , var.
   , toupper(substring(visit.,2,3))
   , summary(pool(with(
     data = mice.full.fit
     , expr = eval(parse(text=paste('lm(I(', var., visit., '-', var., '.w0) \\ ^{\circ} 0 + treat + sex + I(', var., '.w0 - mean(', var., '.w0)))', sep='')))
```

```
)))$estimate[1]
,summary(pool(with(
 data = mice.full.fit
 , expr = eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) ~ 0 + treat + sex + I(', var., '.w0 - mean(', var., '.w0)))', sep='')))
)))$std.error[1]
,summary(pool(with(
 data = mice.full.fit
 , expr = eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) \sim 0 + treat + sex + I(', var., '.w0 - mean(', var., '.w0)))', sep='')))
)))$estimate[2]
,summary(pool(with(
 data = mice.full.fit
```

```
, expr = eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) ~ 0 + treat + sex + I(', var., '.w0 - mean(', var., '.w0)))', sep='')))
)))$std.error[2]
,summary(pool(with(
 data = mice.full.fit
 , expr = eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) \sim 0 + treat + sex + I(', var., '.w0 - mean(', var., '.w0)))', sep='')))
)))$estimate[3]
,summary(pool(with(
 data = mice.full.fit
 , expr = eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) \sim 0 + treat + sex + I(', var., '.w0 - mean(', var., '.w0)))', sep='')))
)))$std.error[3]
,summary(pool(with(
```

```
data = mice.full.fit
 , expr = eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) ~ treat + sex + I(', var., '.w0 - mean(', var., '.w0)))', sep=")))
)))$estimate[1]
,summary(pool(with(
 data = mice.full.fit
 , expr = eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) ~ treat + sex + I(', var., '.w0 - mean(', var., '.w0)))', sep=")))
)))$std.error[1]
,summary(pool(with(
 data = mice.full.fit
 , expr = eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) ~ treat + sex + I(', var., '.w0 - mean(', var., '.w0)))', sep=")))
)))$estimate[2]
```

```
,summary(pool(with(
  data = mice.full.fit
  , expr = eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) ~ treat + sex + I(', var., '.w0 - mean(', var., '.w0)))', sep=")))
 )))$std.error[2]
))
## Include complete case analysis
if (MNAR.type == 1) {
 output <- rbind(output, c(</pre>
  c('CC')
  , 'diff - orig'
  , var.
```

```
, toupper(substring(visit.,2,3))
      , summary(eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) \sim 0 + treat + sex + I(', var., '.w0 - mean(', var., '.w0, na.rm=T)),
data=imp.data)', sep="))))$coef[1,1:2]
      , summary(eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) \sim 0 + treat + sex + I(', var., '.w0 - mean(', var., '.w0, na.rm=T)),
data=imp.data)', sep="))))$coef[2,1:2]
      , summary(eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) \sim 0 + treat + sex + I(', var., '.w0 - mean(', var., '.w0, na.rm=T)),
data=imp.data)', sep="))))$coef[3,1:2]
      , summary(eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) ~ treat + sex + I(', var., '.w0 - mean(', var., '.w0, na.rm=T)),
data=imp.data)', sep="))))$coef[2,1:2]
      , summary(eval(parse(text=paste('lm(I(', var., visit., ' - ', var., '.w0) ~ treat + sex + I(', var., '.w0 - mean(', var., '.w0, na.rm=T)),
data=imp.data)', sep="))))$coef[3,1:2]
    ))
```

```
}; rm(visit.)
 }; rm(var., var.list)
 rm(mice.full.fit)
}; rm(MNAR.type)
output
output <- as.data.frame(output)</pre>
names(output) <- c('analysis', 'type', 'var', 'visit', 'est.C', 'se.C', 'est.A', 'se.A', 'est.B', 'se.B', 'est.BvC', 'se.BvC', 'se.BvC')
for (col. in 5:ncol(output)) output[,col.] <- as.numeric(output[,col.]); rm(col.)
```

